CLINICAL TRIAL: NCT04619719
Title: Multi-Center, Randomized Control Trial to Study the Effectiveness of Hyperbaric Oxygen for COVID-19 Patients With Moderate to Severe Hypoxemia
Brief Title: Hyperbaric Oxygen for COVID-19 Patients With Moderate to Severe Hypoxemia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of patients
Sponsor: Legacy Health System (Other)
Responsible Party: Principal Investigator, Enoch Huang, Principal Investigator, Legacy Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-00897
Record Dates: First submitted 2020-11-05; First posted 2020-11-06 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Covid19
Keywords: Hyperbaric Oxygen
MeSH Terms: conditions — COVID-19 | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Hyperbaric Oxygen (Experimental): Hyperbaric Oxygen Therapy (HBOT) + Standard of Care (SOC) as defined by current best practice treatments for COVID-19
  Interventions: Device: Hyperbaric Oxygen Therapy (HBOT)
- Standard of Care (No Intervention): Standard of Care (SOC) as defined by current best practice treatments for COVID-19

INTERVENTIONS:
Device: Hyperbaric Oxygen Therapy (HBOT) — Patients assigned to the treatment arm will receive up to 5 treatments of hyperbaric oxygen therapy administered daily at 2.0 atmospheres for 90 minutes per session.
  Arms: Hyperbaric Oxygen

SUMMARY:
Of the many treatments proposed for COVID-19, few directly address the severe hypoxia among COVID-19 patients. Interim results from our single-center, non-randomized clinical trial (NCT04332081) suggest that hyperbaric oxygen therapy may reduce inpatient mortality or the need for mechanical ventilation among COVID-19 patients by more than half. Hyperbaric oxygen therapy is delivered by increasing the atmospheric pressure surrounding a patient, which results in increased oxygen delivery to a patient's blood at a rate higher than any other available modality. It is already FDA-approved for several indications, including conditions with impaired gas exchange and severe infectious processes. Furthermore, several studies have found that hyperbaric oxygen therapy inhibits the production of proinflammatory cytokines, which may play a role in the pathophysiology of COVID-19. The goal of this proposal is to perform a multi-center, randomized controlled trial to evaluate the short-term and long-term efficacy of hyperbaric oxygen therapy for COVID-19 patients. This proposal will rigorously test whether hyperbaric oxygen therapy can reduce the substantial mortality and morbidity of this challenging disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Positive COVID 19 test or clear clinical diagnosis of COVID-19. Positive COVID-19 test will be confirmed based on a PCR or antigen test result or patient reported history. Clear clinical diagnosis of COVID-19 will be a combination of respiratory symptoms and clinical findings based on laboratory values and radiographs.
3. Moderate to severe hypoxemia defined by a baseline supplemental oxygen requirement of 6 liters or higher (including high flow oxygenation devices) as measured within the 24 hours before enrollment

Exclusion Criteria:

1. Pregnancy
2. Untreated pneumothorax, which must be evaluated with a baseline chest radiograph or computerized tomography scan at least 72 hours prior to enrollment
3. Presence of pneumomediastinum, pneumopericardium, significant subcutaneous emphysema, or pulmonary blebs, which should also be evaluated with a baseline chest radiograph prior to enrollment
4. Current invasive mechanical ventilation
5. Current non-invasive mechanical ventilation
6. Any patient who will not be stable for transport to the hyperbaric chamber, in addition to any relative contraindications identified by the treating hyperbaric physician or inpatient hospital team (e.g., severely impaired cardiac output due to significant myocardial injury).
7. Any patient without the capacity to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Incidence of 60-Day Patient Mortality | 60 days
  Patient mortality is defined as death from any cause at 60 days after enrollment in the study

SECONDARY OUTCOMES:
Time to Mechanical Ventilation | Duration of inpatient hospitalization, approximately 2 to 4 weeks
Number of Patients with Ongoing Clinical Symptoms | 60 days
  Study participants will be asked about persistent symptoms at 60 days after hospitalization for COVID-19 (i.e., fatigue, dyspnea, joint pain, etc.)
Number of Participants Displaying Presence of Any Pulmonary Function Abnormality | 6 months
  Measured by spirometry and other lung tests (forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), FEV1/FVC, diffusing capacity of the lung for carbon monoxide (DLCO)).
Number of Participants Displaying Presence of Any Pulmonary Function Abnormality | 12 months
  Measured by spirometry and other lung tests (forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), FEV1/FVC, diffusing capacity of the lung for carbon monoxide (DLCO)).

CONTACTS AND LOCATIONS:
Overall Officials: Enoch Huang, MD, Principal Investigator — Legacy Research Institute
Locations (3):
- United States (3):
  - Bozeman Health, Bozeman, Montana
  - NYU Winthrop Hospital, Mineola, New York
  - Legacy Emanuel Medical Center, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to David.Lee@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.